CLINICAL TRIAL: NCT04318873
Title: Evaluation of Demonstrations to End Childhood Hunger - CN DietQual
Acronym: EDECHCNDIETQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USDA Food and Nutrition Service (U.S. Federal Agency)
Collaborators: Mathematica Policy Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AG-3198-C-14-0019 (CN DietQ)
Record Dates: First submitted 2019-12-12; First posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Diet, Healthy
Keywords: Diet quality; Children; Fruit and vegetable voucher; Food box; Nutrition assistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Packed Promise Demonstration Benefits (Experimental): Treatment households (n=2,143) received one food box per eligible child, per month, delivered to the household, which contained (1) shelf-stable foods, including 6 protein-rich items, 2 dairy items, 4 grain foods, 4 cans of fruit, and 12 cans of vegetables; (2) a nutrition education handout (e.g., a recipe); and (3) a $15 Fresh Check for frozen or fresh fruits and vegetables that participants could redeem at any of 38 Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)-authorized stores or farmers' markets in the study counties.
  Interventions: Other: Packed Promise Demonstration Benefits
- Control Group (No Intervention): Control households (n=2,607) did not receive the treatment benefits but still could participate in other available nutrition assistance programs.

INTERVENTIONS:
Other: Packed Promise Demonstration Benefits — Monthly: Home-delivered food box, nutrition education handout, and $15 monthly voucher for fruits and vegetables
  Arms: Packed Promise Demonstration Benefits

SUMMARY:
The 2010 Child Nutrition Reauthorization provided funding to test innovative strategies to end childhood hunger and food insecurity. Demonstration projects were funded in Chickasaw Nation, Kentucky, Navajo Nation, Nevada, and Virginia. This study focuses on Chickasaw Nation and the diet quality of child participants.

School districts were matched, and then one was randomly assigned to either a treatment (n=20) or control group (n=20). Treatment households received one food box per eligible child, per month, delivered to the household, which contained (1) shelf-stable foods, including 6 protein-rich items, 2 dairy items, 4 grain foods, 4 cans of fruit, and 12 cans of vegetables; (2) a nutrition education handout (e.g., a recipe); and (3) a $15 Fresh Check for frozen or fresh fruits and vegetables that participants could redeem at any of 38 Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)-authorized stores or farmers' markets in the study counties. Control households did not receive the treatment benefits but still could participate in other available nutrition assistance programs.

DETAILED DESCRIPTION:
Objective: To reduce childhood food insecurity and hunger, increase families' consumption of nutritious foods, increase the diversity of foods in the home, and ultimately improve diet quality and well-being among children.

Target Population: 40 school districts (115 schools) in 12 counties within the Chickasaw Nation territory in Oklahoma. Within these districts, households with school-age children (both Native American and non-Native American) who were eligible for free school meals or attended a school that participated in the community eligibility provision were eligible to participate in the project.

Intervention School districts were matched, and then one was randomly assigned to either a treatment (n=20) or control group (n=20). Treatment households received one food box per eligible child, per month, delivered to the household, which contained (1) shelf-stable foods, including 6 protein-rich items, 2 dairy items, 4 grain foods, 4 cans of fruit, and 12 cans of vegetables; (2) a nutrition education handout (e.g., a recipe); and (3) a $15 Fresh Check for frozen or fresh fruits and vegetables that participants could redeem at any of 38 Special Supplemental Nutrition Program for Women, Infants, and Children (WIC)-authorized stores or farmers' markets in the study counties. Control households did not receive the treatment benefits but still could participate in other available nutrition assistance programs.

ELIGIBILITY:
Inclusion Criteria:

* 40 school districts (115 schools) in 12 counties within the Chickasaw Nation territory in Oklahoma.
* Within these districts, households with school-age children (both Native American and non-Native American) who were eligible for free National School Lunch Program meals or attended a school that participated in the community eligibility provision were eligible to participate in the project.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 4750 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Daily consumed fruits and vegetables | 30 Days
  The dietary measures used the food frequency questions developed for the 2009-2010 National Health and Nutrition Examination Survey (NHANES) Dietary Screener Questionnaire. For these questions, parents or guardians were asked how often (per day, per week, or per month) a randomly selected child (age 2 or older) in the household consumed food and beverages from 19 categories during the last 30 days.
  The National Cancer Institute's (NCI's) Dietary Screener Questionnaire data processing and scoring procedures were used to convert parent and caregiver reports of their child's daily, weekly, and monthly consumption into standardized daily amounts. Higher scores indicate higher consumption of the food item.
Daily consumed whole grains | 30 Days
  The dietary measures used the food frequency questions developed for the 2009-2010 National Health and Nutrition Examination Survey (NHANES) Dietary Screener Questionnaire. For these questions, parents or guardians were asked how often (per day, per week, or per month) a randomly selected child (age 2 or older) in the household consumed food and beverages from 19 categories during the last 30 days.
  The National Cancer Institute's (NCI's) Dietary Screener Questionnaire data processing and scoring procedures were used to convert parent and caregiver reports of their child's daily, weekly, and monthly consumption into standardized daily amounts. Higher scores indicate higher consumption of the food item.
Daily consumed added sugars | 30 Days
  The dietary measures used the food frequency questions developed for the 2009-2010 National Health and Nutrition Examination Survey (NHANES) Dietary Screener Questionnaire. For these questions, parents or guardians were asked how often (per day, per week, or per month) a randomly selected child (age 2 or older) in the household consumed food and beverages from 19 categories during the last 30 days.
  The National Cancer Institute's (NCI's) Dietary Screener Questionnaire data processing and scoring procedures were used to convert parent and caregiver reports of their child's daily, weekly, and monthly consumption into standardized daily amounts. Higher scores indicate higher consumption of the food item.

SECONDARY OUTCOMES:
Food shopping frequency | 30 Days
  Number of times went food shopping
Type of grocery store used | 30 Days
  Types of grocery stores visited to purchase food
Distance traveled from home to grocery stores | 30 Days
  Distance in miles from home to grocery store where food purchsed
Number of family dinners per week | 30 Days
  Number of family dinners per week

CONTACTS AND LOCATIONS:
Overall Officials: Michael Burke, PhD, Study Director — USDA Food and Nutrition Service

IPD SHARING:
Plan to Share IPD: Yes
Public-use data files are available by request by contacting Michael Burke (michael.burke@usda.gov) or the Office of Policy Support within the USDA Food and Nutrition Service.

REFERENCES:
- [Derived] Cabili C, Briefel R, Forrestal S, Gabor V, Chojnacki G. A Cluster Randomized Controlled Trial of a Home-Delivered Food Box on Children's Diet Quality in the Chickasaw Nation Packed Promise Project. J Acad Nutr Diet. 2021 Jan;121(1S):S59-S69. doi: 10.1016/j.jand.2020.08.012. PMID 33342526
- See also: Final Report — https://www.fns.usda.gov/ops/evaluation-demonstration-projects-ech